CLINICAL TRIAL: NCT02744716
Title: Effects of Aspirin and Intrauterine Balloon on the Post-operative Uterine Endometrial Repair and Reproductive Prognosis in Patients With Severe Intrauterine Adhesion: a Prospective Cohort Study
Brief Title: Effects of Aspirin on Uterine Endometrial Repair Severe Intrauterine Adhesion
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: First Affiliated Hospital, Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Yuqing Chen, Deputy chief physician, First Affiliated Hospital, Sun Yat-Sen University
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: aspirin
Record Dates: First submitted 2016-04-09; First posted 2016-04-20 (Estimated); Last update posted 2016-04-20 (Estimated); Status verified 2016-04

CONDITIONS: Intrauterine Adhesion
Keywords: intrauterine balloon; uterine endometrial repair; intrauterine adhesion; aspirin
MeSH Terms: conditions — Gynatresia | interventions — Aspirin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (3):
- non-balloon group (Experimental): with aspirin
  Interventions: Drug: Aspirin
- balloon group (Experimental): with aspirin and intrauterine balloon
  Interventions: Drug: Aspirin; Device: intrauterine balloon
- control group (No Intervention): without aspirin and intrauterine balloon

INTERVENTIONS:
Drug: Aspirin — low dose of Aspirin after operation
  Other Names: low dose of Aspirin
  Arms: balloon group; non-balloon group
Device: intrauterine balloon — insert intrauterine balloon after operation
  Other Names: Balloon stent
  Arms: balloon group

SUMMARY:
This study aimed To investigate the effects of estrogen in combination with aspirin and intrauterine balloon on the uterine endometrial repair and reproductive prognosis in patients after surgery for severe intrauterine adhesion .

DETAILED DESCRIPTION:
This cohort study was conducted to investigate whether aspirin could promote the endometrial growth and repair, reduce the recurrence of intrauterine adhesion and improve the menstruation and reproductive prognosis after surgery for severe intrauterine adhesion. Menstruation was evaluated for the first time with a method similar to visual analogue scale (VAS) in which the menstruation was assessed by the patients themselves with 0 as amenorrhea and 100 as normal menstruation. This evaluation avoids the vague terms (such as large or small menstrual blood volume) in previous evaluations and considers the individual difference in menstrual blood volume and different understanding about the menstrual blood volume. Thus, this evaluation is easy to master, quantify and analyze.

ELIGIBILITY:
Inclusion Criteria:

* Pre-operative adhesion score was ≥9
* The prior menstrual cycle was regular, and the sex hormone was normal
* Patients had fertility requirement
* Male semen examination showed normal; (5) There were no severe systemic diseases, and no contradictions to aspirin, estrogen and surgery

Exclusion Criteria:

* Pre-operative adhesion score was <9
* Prior menstrual cycle was irregular and sex hormone was abnormal, or patients had endocrine factors that caused amenorrhea, menstrual reduction and infertility
* Patients had no fertility requirement
* Patients had male factor infertility
* Patients had contradictions to estrogen and aspirin such as cancers (breast cancer and endometrial cancer), thrombotic diseases, allergy to antipyretic analgesics, severe liver injury, hypoprothrombinemia, vitamin K deficiency, hemophilia, thrombocytopenia, gastric or duodenal ulcer and asthma.

Ages: 21 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2011-05; Primary Completion 2016-01 (Actual); Study Completion 2016-01 (Actual)

PRIMARY OUTCOMES:
Endometrial Thickness of All Participants in the Mid Menstrual Measured by Color Doppler Ultrasound | Within the first 3 months after surgery

SECONDARY OUTCOMES:
Menstruation Pattern(Improvement or No Significant Change) of All Participants | Within the first 3 months after surgery
  A method similar to VAS was employed for the evaluation of post-operative menstruation with 0 as amenorrhea and 100 as normal menstruation.
Reduction of American Fertility Society adhesion score at Second-look hysteroscopy of All Participants | Within the first 3 months after surgery
  The severity and extent of intrauterine adhesions were scored according to a classification system recommended by the American Fertility Society (AFS) (1988 version) [7]. A score of 1-4 was considered to represent mild adhesions, a score of 5-8 was considered to represent moderate adhesions and a score of 9-12 represented severe adhesions.
Number of Participants With Pregnancy after operation | three years

CONTACTS AND LOCATIONS:
Overall Officials: chen yu qing, Deputy chief, Principal Investigator — First Affiliated Hospital, Sun Yat-Sen University
Locations (1):
- the First Affiliated Hospital of Sun Yat-sen University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Deans R, Abbott J. Review of intrauterine adhesions. J Minim Invasive Gynecol. 2010 Sep-Oct;17(5):555-69. doi: 10.1016/j.jmig.2010.04.016. Epub 2010 Jul 24. PMID 20656564
- [Background] Yang JH, Chen MJ, Chen CD, Chen SU, Ho HN, Yang YS. Optimal waiting period for subsequent fertility treatment after various hysteroscopic surgeries. Fertil Steril. 2013 Jun;99(7):2092-6.e3. doi: 10.1016/j.fertnstert.2013.01.137. Epub 2013 Feb 22. PMID 23433831
- [Background] Sedgh G, Singh S, Henshaw SK, Bankole A. Legal abortion worldwide in 2008: levels and recent trends. Int Perspect Sex Reprod Health. 2011 Jun;37(2):84-94. doi: 10.1363/3708411. PMID 21757423
- [Background] Yu D, Wong YM, Cheong Y, Xia E, Li TC. Asherman syndrome--one century later. Fertil Steril. 2008 Apr;89(4):759-79. doi: 10.1016/j.fertnstert.2008.02.096. PMID 18406834
- [Background] Chen Y, Chang Y, Yao S. Role of angiogenesis in endometrial repair of patients with severe intrauterine adhesion. Int J Clin Exp Pathol. 2013 Jun 15;6(7):1343-50. Print 2013. PMID 23826415
- [Background] Wada I, Hsu CC, Williams G, Macnamee MC, Brinsden PR. The benefits of low-dose aspirin therapy in women with impaired uterine perfusion during assisted conception. Hum Reprod. 1994 Oct;9(10):1954-7. doi: 10.1093/oxfordjournals.humrep.a138366. PMID 7844233
- [Background] Kaandorp SP, Goddijn M, van der Post JA, Hutten BA, Verhoeve HR, Hamulyak K, Mol BW, Folkeringa N, Nahuis M, Papatsonis DN, Buller HR, van der Veen F, Middeldorp S. Aspirin plus heparin or aspirin alone in women with recurrent miscarriage. N Engl J Med. 2010 Apr 29;362(17):1586-96. doi: 10.1056/NEJMoa1000641. Epub 2010 Mar 24. PMID 20335572
- [Background] Lin YH, Jang TN, Hwang JL, Huang LW, Seow KM, Hsieh BC, Huang CH. Bacterial colonization with balloon uterine stent placement in the uterus for 30 days: a randomized controlled clinical trial. Fertil Steril. 2015 Feb;103(2):513-8.e2. doi: 10.1016/j.fertnstert.2014.10.032. Epub 2014 Nov 20. PMID 25467040
- [Background] The American Fertility Society classifications of adnexal adhesions, distal tubal occlusion, tubal occlusion secondary to tubal ligation, tubal pregnancies, mullerian anomalies and intrauterine adhesions. Fertil Steril. 1988 Jun;49(6):944-55. doi: 10.1016/s0015-0282(16)59942-7. No abstract available. PMID 3371491
- [Background] Evans-Hoeker EA, Young SL. Endometrial receptivity and intrauterine adhesive disease. Semin Reprod Med. 2014 Sep;32(5):392-401. doi: 10.1055/s-0034-1376358. Epub 2014 Jun 24. PMID 24959821
- [Background] Lin XN, Zhou F, Wei ML, Yang Y, Li Y, Li TC, Zhang SY. Randomized, controlled trial comparing the efficacy of intrauterine balloon and intrauterine contraceptive device in the prevention of adhesion reformation after hysteroscopic adhesiolysis. Fertil Steril. 2015 Jul;104(1):235-40. doi: 10.1016/j.fertnstert.2015.04.008. Epub 2015 Apr 30. PMID 25936237
- [Background] Bosteels J, Weyers S, Mol BW, D'Hooghe T. Anti-adhesion barrier gels following operative hysteroscopy for treating female infertility: a systematic review and meta-analysis. Gynecol Surg. 2014;11(2):113-127. doi: 10.1007/s10397-014-0832-x. Epub 2014 Mar 14. PMID 24795547
- [Background] Bosteels J, Weyers S, Kasius J, Broekmans FJ, Mol BW, D'Hooghe TM. Anti-adhesion therapy following operative hysteroscopy for treatment of female subfertility. Cochrane Database Syst Rev. 2015 Nov 9;(11):CD011110. doi: 10.1002/14651858.CD011110.pub2. PMID 26559098